CLINICAL TRIAL: NCT04382859
Title: TOTEM: Trial of TAP Block Effective Medications
Acronym: TOTEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Michigan University School of Medicine (Other)
Responsible Party: Principal Investigator, Melinda Abernethy, Associate Professor, Western Michigan University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WMed-2020-0601
Record Dates: First submitted 2020-03-01; First posted 2020-05-11 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP block with liposomal bupivacaine (Active Comparator): Active comparator
  Interventions: Procedure: Transversus abdominis plane (TAP) block with liposomal bupivacaine
- TAP block with 0.25% bupivacaine (Other): Standard comparator
  Interventions: Procedure: Transversus abdominis plane (TAP) block with liposomal bupivacaine

INTERVENTIONS:
Procedure: Transversus abdominis plane (TAP) block with liposomal bupivacaine — Transversus abdominis plane (TAP) blocks are safe and effective procedures for the provision of postoperative pain management following abdominal procedures (3) and have been widely used across specialties with reduction in postoperative pain and narcotic use (4-7).

SUMMARY:
Our goal is to determine if liposomal bupivacaine compared to standard bupivacaine results in increased pain control and decreased narcotic pain medication use when used in TAP blocks prior to laparoscopic hysterectomies for benign indications.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing non robotic assisted laparoscopic surgery for benign gynecologic conditions
* English speaking

Exclusion Criteria:

* Known current malignancy
* Contraindication to medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Pain rating 1 hour post operation | 1 hour post operation
  Participant-reported pain rating on a numeric 0 - 10 scale, with rating of 0 representing no pain and rating 10 representing worst pain
Pain rating 2 hours post operation | 2 hours post operation
  Participant-reported pain rating on a numeric 0 - 10 scale, with rating of 0 representing no pain and rating 10 representing worst pain
Pain rating 4 hours post operation | 4 hours post operation
  Participant-reported pain rating on a numeric 0 - 10 scale, with rating of 0 representing no pain and rating 10 representing worst pain
Pain rating 72 hours post operation | 72 hours post operation
  Participant-reported pain rating on a numeric 0 - 10 scale, with rating of 0 representing no pain and rating 10 representing worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Abernethy, MD, Principal Investigator — Western Michigan University Homer Stryker M.D. School of Medicine
Locations (1):
- Bronson Methodist Hospital, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No